CLINICAL TRIAL: NCT06476210
Title: The Safety and Efficacy of BDL(Bedaquiline Plus Delamanid Plus Linezolid) Regimen in Subjects With Pulmonary Infection of Multi-drug Resistant Tuberculosis (MDR-TB) or Rifampicin-Resistant Tuberculosis (RR-TB)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Collaborators: Public Health Clinical Medical Center of Chengdu (Unknown); Wuhan Institute for Tuberculosis Control (Other); Changsha Central Hospital (Other); Anhui Chest Hospital (Other); Hunan Chest Hospital (Unknown); Shandong Public Health Clinical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YNLX-2024-009
Record Dates: First submitted 2024-06-14; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BDL interventionv group (Experimental)
  Interventions: Drug: BDL regimen

INTERVENTIONS:
Drug: BDL regimen — Drug:bedaquiline 100mg tablets
  Other Names:
  Bdq TMC-207 bedaquiline 400 mg once daily for 2 weeks then 200mg 3 times per week
  Drug:delamanid 50mg tablets
  Other Names:
  Dlm OPC-67683 delamanid 100mg 2 times daily
  Drug:linezolid Scored 600mg tablets
  Other Names:
  Lzd linezolid 600mg once daily

SUMMARY:
The goal of this investigator initiated trial (IIT) is to learn if a 6-9months BDL regimen (bedaquiline plus delamanid plus linezolid）works to treat adults with multi-drug resistant tuberculosis or rifampicin-resistant pulmonary tuberculosis, in the context of Pretomanid not available in China. It will also learn about the safety of BDL regimen.

The main questions it aims to answer are:

1. What is the percentage of participants with favorable treatment outcome at the end of treatment?
2. What are the frequency and degree of AE and SAE associated with BDL regimen?

Participants will take Bedaquiline +Delamanid+ Linezolid for 6 months, option for 9 months for subjects who remain culture positive at month 4 to 6. Safety and efficacy data will be monitored and collected during treatment. A 12 month follow-up will be conducted after treatment completion.

ELIGIBILITY:
Inclusion Criteria

* 1.A patient with multi-drug resistant/rifampicin-resistant pulmonary tuberculosis (MDR/RR-TB) with recent laboratory evidence (culture or molecular testing) within the last two months
* 2.Age 18 years above
* 3.No prior use of neither bedaquiline, delamanid, linezolid, or use for less than 4 weeks
* 4.Positive culture result for mycobacterial at baseline(regardless smear positive or negative). No anti-tuberculosis treatment received within one month.
* 5.For patients who don't have baseline sputum culture results,positive sputum smear and no effective anti-tuberculosis treatment administered
* 6. No history of respiratory failure or heart failure, and no clinically significant manifestations of arrhythmia, with a QTcF under 450ms
* 7.Promise to adhere to the treatment and follow-up schedule, complete treatment monitoring, and promptly report adverse reactions to the responsible physician
* 8.Voluntarily participate in this study and sign the informed consent form

Exclusion Criteria

* 1.According to DMID, peripheral neuropathy is classified as grade 3 or 4. Alternatively, participants with grade 1 or 2 neuropathy, which the investigator believes may progress/worsen during the study
* 2.Elevation of ALT or AST ≥3 times the upper limit of normal, or elevation of total bilirubin and direct bilirubin ≥2 times the upper limit of normal
* 3.Pregnant women or those who intent to pregnant during treatment
* 4.Participants who have participated in other drug trials in the past three months
* 5.Known congenital QT interval prolongation or any disease prolonging the QT interval, or QTc>450 ms
* 6.History of symptomatic arrhythmias or clinically relevant bradycardia
* 7.Any cardiac disease that could precipitate arrhythmias, such as severe hypertension, left ventricular hypertrophy (including hypertrophic cardiomyopathy), or congestive heart failure with decreased left ventricular ejection fraction
* 8.History of known, untreated, persistent hypothyroidism
* 9.Electrolyte disturbances, especially hypokalemia, hypocalcemia, or hypomagnesemia
* 10.History of allergy or known allergic reactions to any investigational drug or related substances
* 11.BMI<17 kg/m2
* 12.Karnofsky performance score under 50, or as determined by the principal investigator, the anticipated survival of the participant is not expected to exceed 6 months
* 13.Participants expected to require surgical intervention following assessment of their pulmonary disease

Withdrawal Criteria

1. Serious adverse events caused by the intervention
2. Confirmed QTcF interval ≥ 500ms or clinically significant ventricular arrhythmias
3. The expert panel deems the continuation of this combination regimen inappropriate
4. The patient requests withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The efficacy outcome at the end of treatment | Baseline (within 9 days before treatment initiation), weeks 1, 2, 4, 6, 8 of treatment, thereafter every 4 weeks until week 26(or 39 weeks for patients require prolonged treatment) during the intervention
  The efficacy outcome of treatment: bacteriological positive patients completed the prescribed treatment course, demonstrating bacteriological response without evidence of treatment failure Notes: bacteriological outcome response:bacterial culture conversion to negative and no recurrence of positivity thereafter Bacteriological conversion refers to confirmed tuberculosis patients having two or more consecutive negative sputum culture results, with at least a 7-day interval between each Recurrence of positivity refers to two or more consecutive sputum cultures were positive after bacteriological conversion, with at least a 7-day interval between each
Frequency of any adverse events (AEs) and serious adverse events (SAEs) occurring during the treatment period | Baseline (within 9 days before treatment initiation), weeks 1-16, 20 and 26 during the intervention

SECONDARY OUTCOMES:
Incidence of patients have bacterial recurrence within 12 months after treatment completion | 3,6,9,12 months after the intervention
Time for sputum culture conversion to stable negativity during treatment | 3,6,9,12 months after the intervention
Proportion of patients who discontinued treatment due to adverse reactions or permanently unable to take the medication | during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Liu, Ph.D, Principal Investigator — Beijing Chest Hostal; Mengqiu Gao, Ph.D, Principal Investigator — Beijing Chest Hospital
Locations (7):
- China (7):
  - Anhui Chest Hospital, Hefei, Anhui
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Wuhan Institute for Tuberculosis Control, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Chest Hospital, Changsha, Hunan
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Public Health Clinical Meadical Center of Chengdu, Chengdu, Sichuan

REFERENCES:
- [Background] Dooley KE, Rosenkranz SL, Conradie F, Moran L, Hafner R, von Groote-Bidlingmaier F, Lama JR, Shenje J, De Los Rios J, Comins K, Morganroth J, Diacon AH, Cramer YS, Donahue K, Maartens G; AIDS Clinical Trials Group (ACTG) A5343 DELIBERATE Study Team. QT effects of bedaquiline, delamanid, or both in patients with rifampicin-resistant tuberculosis: a phase 2, open-label, randomised, controlled trial. Lancet Infect Dis. 2021 Jul;21(7):975-983. doi: 10.1016/S1473-3099(20)30770-2. Epub 2021 Feb 12. PMID 33587897
- [Background] Lachatre M, Rioux C, Le Du D, Frechet-Jachym M, Veziris N, Bouvet E, Yazdanpanah Y. Bedaquiline plus delamanid for XDR tuberculosis. Lancet Infect Dis. 2016 Mar;16(3):294. doi: 10.1016/S1473-3099(16)00047-5. No abstract available. PMID 26973310
- [Background] Kim CT, Kim TO, Shin HJ, Ko YC, Hun Choe Y, Kim HR, Kwon YS. Bedaquiline and delamanid for the treatment of multidrug-resistant tuberculosis: a multicentre cohort study in Korea. Eur Respir J. 2018 Mar 22;51(3):1702467. doi: 10.1183/13993003.02467-2017. Print 2018 Mar. PMID 29545276
- [Background] Gao JT, Du J, Wu GH, Pei Y, Gao MQ, Martinez L, Fan L, Chen W, Xie L, Chen Y, Wang H, Jin L, Li GB, Zong PL, Xiong Y, Wu QH, Li MW, Yan XF, Miao YF, Cai QS, Li XJ, Bai DP, Geng SJ, Yang GL, Tang PJ, Zeng Y, Chen XH, Li TX, Cai C, Zhou Y, Zhuo M, Wang JY, Guan WL, Xu L, Shi JC, Shu W, Cheng LL, Teng F, Ning YJ, Xie SH, Sun YX, Zhang LJ, Liu YH. Bedaquiline-containing regimens in patients with pulmonary multidrug-resistant tuberculosis in China: focus on the safety. Infect Dis Poverty. 2021 Mar 19;10(1):32. doi: 10.1186/s40249-021-00819-2. PMID 33736710
- [Background] Blair HA, Scott LJ. Delamanid: a review of its use in patients with multidrug-resistant tuberculosis. Drugs. 2015 Jan;75(1):91-100. doi: 10.1007/s40265-014-0331-4. PMID 25404020
- [Background] Pieterman ED, Keutzer L, van der Meijden A, van den Berg S, Wang H, Zimmerman MD, Simonsson USH, Bax HI, de Steenwinkel JEM. Superior Efficacy of a Bedaquiline, Delamanid, and Linezolid Combination Regimen in a Mouse Tuberculosis Model. J Infect Dis. 2021 Sep 17;224(6):1039-1047. doi: 10.1093/infdis/jiab043. PMID 33502537
- [Background] Tasneen R, Williams K, Amoabeng O, Minkowski A, Mdluli KE, Upton AM, Nuermberger EL. Contribution of the nitroimidazoles PA-824 and TBA-354 to the activity of novel regimens in murine models of tuberculosis. Antimicrob Agents Chemother. 2015 Jan;59(1):129-35. doi: 10.1128/AAC.03822-14. Epub 2014 Oct 20. PMID 25331697
- [Background] Upton AM, Cho S, Yang TJ, Kim Y, Wang Y, Lu Y, Wang B, Xu J, Mdluli K, Ma Z, Franzblau SG. In vitro and in vivo activities of the nitroimidazole TBA-354 against Mycobacterium tuberculosis. Antimicrob Agents Chemother. 2015 Jan;59(1):136-44. doi: 10.1128/AAC.03823-14. Epub 2014 Oct 20. PMID 25331696
- [Background] Matsumoto M, Hashizume H, Tomishige T, Kawasaki M, Tsubouchi H, Sasaki H, Shimokawa Y, Komatsu M. OPC-67683, a nitro-dihydro-imidazooxazole derivative with promising action against tuberculosis in vitro and in mice. PLoS Med. 2006 Nov;3(11):e466. doi: 10.1371/journal.pmed.0030466. PMID 17132069
- [Background] Zhang F, Li S, Wen S, Zhang T, Shang Y, Huo F, Xue Y, Li L, Pang Y. Comparison of in vitro Susceptibility of Mycobacteria Against PA-824 to Identify Key Residues of Ddn, the Deazoflavin-Dependent Nitroreductase from Mycobacterium tuberculosis. Infect Drug Resist. 2020 Mar 11;13:815-822. doi: 10.2147/IDR.S240716. eCollection 2020. PMID 32210596
- [Background] Stinson K, Kurepina N, Venter A, Fujiwara M, Kawasaki M, Timm J, Shashkina E, Kreiswirth BN, Liu Y, Matsumoto M, Geiter L. MIC of Delamanid (OPC-67683) against Mycobacterium tuberculosis Clinical Isolates and a Proposed Critical Concentration. Antimicrob Agents Chemother. 2016 May 23;60(6):3316-22. doi: 10.1128/AAC.03014-15. Print 2016 Jun. PMID 26976868
- [Background] Keller PM, Homke R, Ritter C, Valsesia G, Bloemberg GV, Bottger EC. Determination of MIC distribution and epidemiological cutoff values for bedaquiline and delamanid in Mycobacterium tuberculosis using the MGIT 960 system equipped with TB eXiST. Antimicrob Agents Chemother. 2015 Jul;59(7):4352-5. doi: 10.1128/AAC.00614-15. Epub 2015 May 4. PMID 25941226
- [Background] Liu Y, Matsumoto M, Ishida H, Ohguro K, Yoshitake M, Gupta R, Geiter L, Hafkin J. Delamanid: From discovery to its use for pulmonary multidrug-resistant tuberculosis (MDR-TB). Tuberculosis (Edinb). 2018 Jul;111:20-30. doi: 10.1016/j.tube.2018.04.008. Epub 2018 May 3. PMID 30029909
- [Background] Conradie F, Diacon AH, Ngubane N, Howell P, Everitt D, Crook AM, Mendel CM, Egizi E, Moreira J, Timm J, McHugh TD, Wills GH, Bateson A, Hunt R, Van Niekerk C, Li M, Olugbosi M, Spigelman M; Nix-TB Trial Team. Treatment of Highly Drug-Resistant Pulmonary Tuberculosis. N Engl J Med. 2020 Mar 5;382(10):893-902. doi: 10.1056/NEJMoa1901814. PMID 32130813
- [Background] Trebucq A, Schwoebel V, Kashongwe Z, Bakayoko A, Kuaban C, Noeske J, Hassane S, Souleymane B, Piubello A, Ciza F, Fikouma V, Gasana M, Ouedraogo M, Gninafon M, Van Deun A, Cirillo DM, Koura KG, Rieder HL. Treatment outcome with a short multidrug-resistant tuberculosis regimen in nine African countries. Int J Tuberc Lung Dis. 2018 Jan 1;22(1):17-25. doi: 10.5588/ijtld.17.0498. Epub 2017 Nov 17. PMID 29149917